CLINICAL TRIAL: NCT03940703
Title: A Phase II, Two-arm Study to Investigate Tepotinib Combined With Osimertinib in MET Amplified, Advanced or Metastatic NSCLC Harboring Activating EGFR Mutations and Having Acquired Resistance to Prior Osimertinib Therapy (INSIGHT 2)
Brief Title: A Study of Tepotinib Plus Osimertinib in Osimertinib Relapsed MET Amplified NSCLC (INSIGHT 2)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MS200095_0031; 2019-001538-33 (EudraCT Number); 2024-512005-87-00 (EU CTIS Number)
Record Dates: First submitted 2019-05-06; First posted 2019-05-07 (Actual); Results first posted 2024-06-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Tepotinib; Osimertinib; Non-Small Cell Lung Cancer; INSIGHT 2; MET amplified
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tepotinib; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tepotinib and Osimertinib (Experimental): Participants received a single oral dose of Tepotinib 500 milligrams (mg) followed by Omisertinib 80 mg once daily until disease progression, death, adverse event leading to discontinuation, study withdrawal or consent withdrawal.
  Interventions: Drug: Tepotinib; Drug: Osimertinib
- Tepotinib Mono-therapy (Experimental): Participants received a single oral dose of Tepotinib 500 mg until disease progression, death, adverse event leading to discontinuation, study withdrawal or consent withdrawal.
  Interventions: Drug: Tepotinib

INTERVENTIONS:
Drug: Tepotinib — Participants were administered with Tepotinib orally once daily at a dose of 500 mg.
Drug: Osimertinib — Participants received Osimertinib at a dose of 80 mg orally once daily.
  Other Names: Tagrisso®
  Arms: Tepotinib and Osimertinib

SUMMARY:
This study was to assess the antitumor activity, safety, tolerability, and pharmacokinetics (PK) of the Mesenchymal-epithelial Transition Factor (MET) inhibitor tepotinib combined with the 3rd generation EGFR inhibitor osimertinib in participants with advanced or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic Non-small Cell Lung Cancer (NSCLC) histology (confirmed by either histology or cytology) with documented activating Epidermal Growth Factor Receptor (EGFR) mutation
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 and a minimum life expectancy of 12 weeks
* Acquired resistance on previous first-line osimertinib. Participants must meet both of the following 2 criteria:
* Radiological documentation of disease progression on first-line osimertinib
* Objective clinical benefit documented during previous osimertinib therapy, defined by either partial or complete radiological response, or durable stable disease (SD) (SD should last greater than (>) 6 months after initiation of osimertinib
* Have received only first-line osimertinib as a prior line of therapy in the non curative advanced or metastatic NSCLC setting
* MET amplification as determined by either FISH testing (central or local) on tumor tissue (TBx) or central blood-based next generation sequencing (LBx). Tumor and blood samples must be collected following progression on prior first-line osimertinib at Prescreening
* Submission of tumor tissue and blood sample obtained after progression on first-line osimertinib, is mandatory for all patients for MET amplification testing
* Submission of tumor tissue during Prescreening or Screening is mandatory for patients with tumor tissue tested by local FISH, to confirm MET amplification status. Central confirmation is not mandated prior to the start of study treatment
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Spinal cord compression or brain metastasis unless asymptomatic, stable or not requiring steroids for at least 2 weeks prior to start of study intervention
* Any unresolved toxicity Grade 2 or more according to National cancer institute common terminology criteria for adverse events( NCI-CTCAE) version 5, from previous anticancer therapy with the exception of alopecia
* Inadequate hematological, liver and renal function
* Impaired cardiac function
* History of interstitial lung disease(ILD) or interstitial pneumonitis including radiation pneumonitis that required steroid treatment
* Hypertension uncontrolled by standard therapies (not stabilized to < 150/90 millimeter of mercury (mmHg)
* Contraindication to the administration of osimertinib
* Other protocol defined exclusion criteria could apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2026-05-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (179):
- United States (49):
  - Yuma Regional Medical Center, Yuma, Arizona
  - Compassionate Care Research Group Inc - Edinger Medical Group, Inc., Fountain Valley, California
  - Memorial Care, Long Beach, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Innovative Clinical Research Institute, Whittier, California
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Holy Cross, Fort Lauderdale, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Ocala Oncology, Ocala, Florida
  - University Cancer and Blood Center, Athens, Georgia
  - Hawaii Cancer Care, Honolulu, Hawaii
  - University of Chicago Medical Center, Chicago, Illinois
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Community Health Network, Indianapolis, Indiana
  - Beacon Health, South Bend, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Pontchartrain, Hammond, Louisiana
  - Medstar Franklin Square Clinical Research Center, Baltimore, Maryland
  - The Center for Cancer & Blood Disorders - Maryland, Bethesda, Maryland
  - Frederick Health- James M Stockman Cancer Institute, Frederick, Maryland
  - Boston Medical Center - Dept. Hematology/Oncology, Boston, Massachusetts
  - Southcoast Center for Cancer Care, Fairhaven, Massachusetts
  - Sparrow Hospital Herbert - Herman Cancer Center, Lansing, Michigan
  - Central Care Cancer Center (CCCC), Bolivar, Missouri
  - St. Louis Cancer Care, LLP, Bridgeton, Missouri
  - Mosaic Life Care, Saint Joseph, Missouri
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - New Jersey Cancer Care and Blood Disorders, Belleville, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - NYU Langone Clinical Cancer Center - NYU Langone Medical Center, New York, New York
  - NYU Langone Clinical Cancer Center - NYU Langone Medical Cente, New York, New York
  - Weill Cornell Medical College - Gastroenterology, New York, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - University Hospitals Seidman, Cleveland, Ohio
  - OhioHealth, Columbus, Ohio
  - Oklahoma Cancer Specialists and Research Institute, Tulsa, Oklahoma
  - Oregon Oncology Specialists, Salem, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Sanford Health, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baptist Cancer Center, Memphis, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Mary Crowley Cancer Research, Dallas, Texas
  - University of Texas MD Anderson Cancer Center - Unit 432 Thoracic Head and Neck Medical Oncology, Houston, Texas
  - Community Cancer Trials of Utah, Ogden, Utah
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Hematology Oncology Associates of Fredericksburg, Fredericksburg, Virginia
  - Northwest Medical Specialties, Tacoma, Washington
- Belgium (3):
  - UZ Antwerpen - Department of Oncology, Edegem
  - UZ Leuven, Gasthuisberg
  - AZ Delta, Roeselare
- China (21):
  - Beijing Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Cancer Hospital, Beijing
  - Jilin Cancer Hospital - Oncology, Changchun
  - The First Hospital of Jilin University, Changchun
  - Hunan Cancer Hospital, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Guangdong General Hospital, Guangzhou
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Affiliated Tumor Hospital of Harbin Medical University, Harbin
  - Anhui Chest Hospital, Hefei
  - Linyi Tumor Hospital, Linyi
  - Jiangsu Province Hospital, Nanjing
  - Shanghai Cancer Hospital, Fudan University, Shanghai
  - Shanghai Chest Hospital, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - The Affiliated Cancer Hospital of Xinjiang Medical university, Ürümqi
  - Hubei Cancer Hospital, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
- France (9):
  - Centre Francois Baclesse - Service d'Oncologie Medicale, Caen
  - Centre Hospitalier Intercommunal de Créteil - Service de Pneumologie, Créteil
  - CHU Limoges - Hôpital Dupuytren - Unite d'Oncologie Thoracique et Cutanée, Limoges
  - Centre Léon Bérard, Lyon
  - Hopital Albert Calmette - CHU Lille - service de pneumologie et immuno allergologie, Nord
  - Hopital Tenon - service pneumologie, Paris
  - Hospital Cochin Service, Service de Pneumologie et Mucoviscidose, Paris
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - Maison du Ha, Pessac
  - CHU de Toulouse - Hôpital Larrey - Service de Pneumologie et Oncologie Pneumologique, Toulouse
- Germany (13):
  - Universitaetsklinikum Koeln - Innere Medizin I, Onkologie, Haematologie, Cologne
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Asklepios Fachkliniken Muenchen-Gauting - Abteilung internistische Onkologie, Gauting
  - Universitaetsklinikum Giessen und Marburg GmbH Standort Giessen, Giessen
  - Universitaetsmedizin Goettingen, Göttingen
  - Evangelisches Krankenhaus Hamm gGmbH, Hamm
  - Evangelisches Krankenhaus Hamm GmbH, Hamm
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - Staedtisches Krankenhaus Kiel, Kiel
  - POIS Leipzig GbR, Leipzig
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
  - Pius-Hospital Oldenburg - Klinik f. Haematologie und Onkologie, Oldenburg
  - Missionsärztliche Klinik, Würzburg
- Hong Kong (3):
  - Queen Elizabeth Hospital - Department of Medicine, Hong Kong
  - The University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong - Emergency Medicine, Shatin
- Italy (11):
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - UOC Oncologia Medica, Lazio
  - IEO Istituto Europeo di Oncologia, Milan
  - Azienda Socio Sanitaria Territoriale di Monza (Presidio San Gerardo) - U.O Oncologia Medica, Monza
  - Ospedale Monaldi, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS - Oncologia Medica 2, Padua
  - AO Ospedali Riuniti Cervello - Presidio Villa Sofia - U.O.S. di Neuroimmunologia, Palermo
  - Azienda Ospedaliero Universitaria Pisana - U.O. Pneumologia II, Pisa
  - Istituto Nazionale Tumori Regina Elena IRCCS - S.C. Oncologia Medica B, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Socio Sanitaria Territoriale Sette Laghi (Presidio Ospedale di Circolo e Fondazione Macchi) - Oncologia Medica, Varese
  - Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma) - U.O.C. Oncologia, Verona
- Japan (11):
  - Hamamatsu University School of Medicine, University Hospital - Dept of Respiratory Medicine, Hamamatsu
  - Saitama Cancer Center, Kitaadachi-gun
  - Kurume University Hospital, Kurume-shi
  - Nagoya University Hospital - Dept of Respiratory Medicine, Nagoya
  - Niigata Cancer Center Hospital - Dept of Internal Medicine, Niigata
  - Hyogo College of Medicine Hospital - Dept of Respiratory Medicine, Nishinomiya-shi
  - Okayama University Hospital - Dept of Respiratory Medicine/Allergy, Okayama
  - Osaka City General Hospital, Osaka
  - Kindai University Hospital, Osakasayama-shi
  - NHO Yamaguchi - Ube Medical Center, Ube-shi
  - Kanagawa Cancer Center - Dept of Respiratory Medicine, Yokohama
- Malaysia (7):
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Beacon International Specialist Centre Sdn Bhd, Kuala Selangor
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Hospital Umum Sarawak, Kuching
  - Sunway Medical Centre, Petaling Jaya, Selangor
  - Hospital Pulau Pinang - Clinic Respiratory, Pulau Pinang
- Netherlands (3):
  - The Netherlands Cancer Institute, Amsterdam
  - Universitair Medisch Centrum Groningen - Department of Internal Medicine, Groningen
  - Maastricht University Medical Center - Dept of Medical Oncology, Maastricht
- Russia (7):
  - SBHI "Krasnoyarsk Regional Oncology Dispensary n.a. A.I. Kryzhanovsky", Krasnoyarsk
  - "VitaMed" LLC, Moscow
  - LLC "Tonus", Nizniy Novgorod
  - BHI of Omsk region "Clinical Oncology Dispensary", Omsk
  - LLC "ClinicaUZI4D", Pyatigorsk
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University - Research Institute of Pulmunology, Saint Petersburg
- Singapore (3):
  - Icon Cancer Centre, Connexion
  - National Cancer Centre - Medical Oncology Pharmacy, Singapore
  - Tan Tock Seng Hospital - CTRU/OCS, Research, Singapore
- South Korea (9):
  - National Cancer Center, Goyang-si
  - Chonnam National University Hwasun Hospital, Hwasun-gun
  - Seoul National University Bundang Hospital, Seongnam-si
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (13):
  - ICO Badalona - Hospital Germans Trias i Pujol - Servicio de Oncologia Medica, Badalona
  - Hospital del Mar - Servicio de Oncologia, Barcelona
  - Hospital Universitari Dexeus - Servicio de Oncologia Medica, Barcelona
  - Hospital Universitari Quiron Dexeus - Servicio de Oncologia Medica, Barcelona
  - Hospital Universitari Vall d'Hebron - Dept of Oncology, Barcelona
  - ICO l´Hospitalet - Hospital Duran i Reynals - Servicio de Oncologia, L'Hospitalet de Llobregat
  - Hospital Universitario Materno-Infantil de Canarias - Servicio de Oncologia, Las Palmas de Gran Canaria
  - Hospital Universitario HM Madrid Sanchinarro - Servicio de Oncologia, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitari Son Espases - Servicio de Oncologia Medica, Palma
  - Hospital Universitario Quiron Madrid - Unidad Integral de Oncologia, Pozuelo de Alarcón
  - Hospital Universitario Virgen Macarena - Servicio de Oncologia, Seville
  - Hospital Universitari i Politecnic La Fe - Servicio de Oncologia Medica, Valencia
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Liou Ying, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
- Thailand (4):
  - Siriraj Hospital, Bangkoknoi
  - Songklanagarind Hospital, Hat Yai
  - Maharaj Nakorn Chiang Mai Hospital, Muang
  - King Chulalongkorn Memorial Hospital, Pathumwan
- Vietnam (6):
  - Bach Mai Hospital, Hanoi
  - K Hospital, Hanoi
  - National Lungs Hospital, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City
  - HCMC Oncology Hospital, Ho Chi Minh City
  - Pham Ngoc Thach Hospital, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Background] F Smit E, Dooms C, Raskin J, Nadal E, Tho LM, Le X, Mazieres J, S Hin H, Morise M, W Zhu V, Tan D, H Holmberg K, Ellers-Lenz B, Adrian S, Brutlach S, Schumacher KM, Karachaliou N, Wu YL. INSIGHT 2: a phase II study of tepotinib plus osimertinib in MET-amplified NSCLC and first-line osimertinib resistance. Future Oncol. 2022 Mar;18(9):1039-1054. doi: 10.2217/fon-2021-1406. Epub 2021 Dec 17. PMID 34918545
- [Derived] Wu YL, Guarneri V, Voon PJ, Lim BK, Yang JJ, Wislez M, Huang C, Liam CK, Mazieres J, Tho LM, Hayashi H, Nhung NV, Chia PL, de Marinis F, Raskin J, Zhou Q, Finocchiaro G, Le AT, Wang J, Dooms C, Kato T, Nadal E, Hin HS, Smit EF, Wermke M, Tan D, Morise M, O'Brate A, Adrian S, Pfeiffer BM, Stroh C, Juraeva D, Strotmann R, Goteti K, Berghoff K, Ellers-Lenz B, Karachaliou N, Le X, Kim TM; INSIGHT 2 investigators. Tepotinib plus osimertinib in patients with EGFR-mutated non-small-cell lung cancer with MET amplification following progression on first-line osimertinib (INSIGHT 2): a multicentre, open-label, phase 2 trial. Lancet Oncol. 2024 Aug;25(8):989-1002. doi: 10.1016/S1470-2045(24)00270-5. PMID 39089305
- [Derived] Hallick J, Baird AM, Falchook G, Le X, Hong D, Viteri S, Raskin J, Reinmuth N, Vlassak S, Militaru M, Paik PK. Plain language summary of the development of tepotinib: a treatment for a subtype of non-small cell lung cancer called MET exon 14 skipping. Future Oncol. 2023 Mar;19(10):683-696. doi: 10.2217/fon-2022-1035. Epub 2023 Mar 31. PMID 36999526
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS200095_0031
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: Targeting MET Clinical Trial Program — https://www.clinicaltrials.targeting-met.com/en

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tepotinib and Osimertinib | Tepotinib Mono-therapy
Started | 128 | 12
Full Analysis Set (FAS) (FAS included all participants who were administered any dose of any study treatment.) | 128 | 12
Safety (SAF) Analysis Set (SAF analysis set included all participants who were administered any dose of any study treatment.) | 128 | 12
Modified Full Analysis Set (mFAS) (mFAS: All FAS/SAF participants who started study treatment on or before the 08 July 2022 (that is [i.e.] date of completion of global enrollment), tested positive for MET amplification by either central test on tumor tissue or liquid biopsy or both, and progressed on first-line osimertinib as the only prior line of therapy in the noncurative advanced or metastatic NSCLC setting. T+ participants also belong to the Primary Analysis Set for Efficacy.) | 105 | 12
Safety run-in Analysis Set (SRIAS) (SRIAS included all FAS/SAF participants treated during the safety run-in period who received at least 75 percent (% )of the tepotinib and osimertinib planned dose and completed the Dose-Limiting Toxicity (DLT) period (3 weeks after start of study treatment), or who experienced a DLT during the DLT period regardless of the received amount of each study treatment component.) | 9 | 0
Pharmacokinetic (PK) Analysis Set (PK analysis set included all FAS/SAF participants who have no important events affecting PK and provide at least one measurable post-dose concentration.) | 120 | 11
Completed | 97 | 12
Not Completed | 31 | 0
Not completed — Still under treatment | 31 | 0

BASELINE CHARACTERISTICS:
Population: Safety (SAF) analysis set included all participants who were administered any dose of any study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tepotinib and Osimertinib | Tepotinib Mono-therapy | Total
Number analyzed (Participants) | 128 | 12 | 140
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59 (10.8) | 61 (9.7) | 60 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 9 | 83
  Male | 54 | 3 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity-Hispanic or Latino | 3 | 0 | 3
  Ethnicity-Not Hispanic or Latino | 124 | 12 | 136
  Ethnicity-Unknown or Not Reported | 1 | 0 | 1
  Race-Asian | 79 | 6 | 85
  Race-Black or African American | 1 | 0 | 1
  Race-Not Collected At This Site | 4 | 2 | 6
  Race-Other | 1 | 0 | 1
  Race-White | 43 | 4 | 47

OUTCOME MEASURES:

1. Primary Outcome: Combined Therapy (Tepotinib+Osimertinib): Number of Participants Experiencing Dose-Limiting Toxicities (DLTs) According to National Cancer Institute Common Terminology Criteria for Adverse Events Version (NCI-CTCAE v 5.0)
Description: DLTs are defined as any of the following toxicities and judged by the Investigator and/or the Sponsor to be not attributable to the disease or disease-related processes under investigation: Grade 4 neutropenia for more than 7 days; Grade greater than or equal to (>=) 3 febrile neutropenia; Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with non-traumatic bleeding; Grade >= 3 nausea/vomiting and/or diarrhea that has not improved within 72 hours despite adequate and optimal treatment; Any other Grade >= 3 non-hematological AE, except alopecia or Grade 3 nauseas/vomiting and/or diarrhea that has improved within 72 hours with optimal treatment.
Time Frame: Up to Day 21 of Cycle 1 (each Cycle is of 21 days)
Population: Safety run-in analysis set (SRIAS): all FAS/SAF participants treated during the safety run-in period who received at least 75% of the tepotinib and osimertinib planned dose and completed the DLT period (3 weeks after start of study treatment), or who experienced a DLT during the DLT period regardless of the received amount of each study treatment component.
Measure: Count of Participants; unit: Participants
Groups:
- Tepotinib + Osimertinib: Participants received 500 milligrams (mg) of tepotinib orally once daily in combination with Osimertinib at a dose of 80 mg orally once daily until disease progression, death, adverse event leading to discontinuation, study withdrawal or consent withdrawal.
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 9
Participants | 1

2. Primary Outcome: Combined Therapy: Objective Response According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1as Per Independent Review Committee in Participants With MET Amplification Determined Centrally by Fluorescence in Situ Hybridization(FISH)
Description: Objective response was defined as percentage of participants with either a confirmed complete response (CR) or partial response (PR) from first administration of study treatment to first observation of progressive disease (PD) .CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: The primary analysis set for efficacy included all mFAS participants with advanced or metastatic Epidermal Growth Factor Receptor mutation positive (EGFRm+) Non-Small Cell Lung Cancer (NSCLC) and Mesenchymal-Epithelial Transition factor (MET) amplification, determined centrally by FISH (central TBx FISH testing [T+]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
percentage of participants | 50.0 [39.7 to 60.3]

3. Secondary Outcome: Combined Therapy: Objective Response According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1as Per Independent Review Committee in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: as for outcome 2
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: The secondary analysis set for efficacy included all modified Full Analysis Set (mFAS) participants with advanced or metastatic Epidermal Growth Factor Receptor mutation positive (EGFRm+) Non-Small Cell Lung Cancer (NSCLC) and Mesenchymal-Epithelial Transition factor (MET) amplification, determined centrally by liquid biopsy (LBx) test (L+).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
percentage of participants | 54.8 [36.0 to 72.7]

4. Secondary Outcome: Monotherapy (Tepotinib): Objective Response According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1 as Per Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 2
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: The primary analysis set for efficacy included all mFAS participants with advanced or metastatic EGFRm+ NSCLC and MET amplification, determined centrally by FISH (central TBx FISH testing [T+]).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Tepotinib Monotherapy: Participants received 500 milligrams (mg) of tepotinib orally once daily until disease progression, death, adverse event leading to discontinuation, study withdrawal or consent withdrawal.
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 12
percentage of participants | 8.3 [0.2 to 38.5]

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment-Related TEAEs
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether considered related to the study intervention or not. A serious AE was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. TEAEs were defined as events with onset date or worsening during the on-treatment period. TEAEs included both serious and non-serious TEAEs. Treatment-related TEAEs is defined as reasonably related to the study intervention.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: Safety (SAF) analysis set included all participants who were administered any dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib | Tepotinib Monotherapy
Number analyzed (Participants) | 128 | 12
Participants
  TEAEs | 126 | 12
  Treatment-related TEAEs | 113 | 9

6. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Laboratory Values Reported as Treatment Related TEAEs
Description: The laboratory measurements included hematology, biochemistry, coagulation and urinalysis. Number of participants with clinically significant abnormalities in laboratory values reported as treatment related TEAEs were reported. Clinical significance was decided by investigator.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: Safety (SAF) analysis set included all participants who were administered any dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib | Tepotinib Monotherapy
Number analyzed (Participants) | 128 | 12
Participants
  Anemia | 2 | 0
  Febrile neutropenia | 1 | 0
  Leukopenia | 1 | 0
  Myelosuppression | 1 | 0
  Neutropenia | 1 | 0
  Lymphocyte count decreased | 1 | 0
  Neutrophil count decreased | 2 | 0
  Platelet count decreased | 3 | 0
  White blood cell count decreased | 3 | 0
  Alanine aminotransferase increased | 2 | 0
  Alkaline phosphatase increased | 1 | 0
  Lipase increased | 3 | 0
  Hypoalbuminemia | 1 | 0
  Urinary tract infection | 0 | 0
  Activated partial thromboplastin time | 0 | 0
  Prothrombin international normalized ratio | 0 | 0

7. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Sign Measurements
Description: Vital signs included systolic blood pressure (SBP) and diastolic blood pressure (DBP), pulse rate (PR), respiratory rate (RR) body weight (BW) and body temperature (BT). Markedly abnormal value (MAV) criteria for vital signs: SBP and DBP: maximal on treatment (TR) increase or decrease greater than (>) 40 millimeter of mercury (mmHg); PR: maximal on TR increase or decrease >40 beats per minute (bpm); RR: maximal on TR increase or decrease >10 breaths per minute (breaths/minute), BW: maximum on TR increase or decrease >=10% and BT: maximal on TR increase greater than or equal to (>=)2 degree Celsius. Number of participants who met the MAV criteria for vital signs at least once post dose were reported.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: Safety (SAF) analysis set included all participants who were administered any dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib | Tepotinib Monotherapy
Number analyzed (Participants) | 128 | 12
Participants
  SBP: maximum on TR increase of >40 mmHg | 2 | 0
  SBP: maximum on TR decrease of >40 mmHg | 6 | 0
  DBP: maximum on TR increase of >40 mmHg | 0 | 0
  DBP: maximum on TR decrease of >40 mmHg | 1 | 0
  RR: maximum on TR increase of >10 beats/min | 1 | 0
  RR: maximum on TR decrease of >10 beats/min | 0 | 0
  PR: maximum on TR increase of > 40 bpm | 4 | 0
  PR: maximum on TR decrease of >40 bpm | 2 | 1
  BW: maximum on TR increase of >=10% | 14 | 1
  BW: maximum on TR decrease of >=10% | 13 | 2
  BT: maximal on TR increase >=2 degree Celsius | 1 | 1

8. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance: Baseline Score Versus (Vs) Worst Post-baseline Score
Description: ECOG performance status measured to assess participant's performance status on a scale of 0 to 5, where 0 = Fully active, able to carry on all pre-disease activities without restriction; 1 = Restricted in physically strenuous activity, ambulatory and able to carry out light or sedentary work; 2 = Ambulatory and capable of all selfcare but unable to carry out any work activities; 3 = Capable of only limited self-care, confined to bed/chair for more than 50 percent of waking hours; 4 = Completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5 = dead. ECOG performance status was reported in terms of number of participants with shifts in score from baseline value vs worst post-baseline value (that is [i.e.] highest score).
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: Safety (SAF) analysis set included all participants who were administered any dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib | Tepotinib Monotherapy
Number analyzed (Participants) | 128 | 12
Participants
  Maximum Baseline score 0, worst post-baseline score 0 | 14 | 3
  Maximum Baseline score 0, worst post-baseline score 1 | 16 | 1
  Maximum Baseline score 0, worst post-baseline score 2 | 3 | 0
  Maximum Baseline score 0, worst post-baseline score 3 | 2 | 0
  Maximum Baseline score 0, worst post-baseline score 4 | 0 | 0
  Maximum Baseline score 0, worst post-baseline score 5 | 0 | 0
  Maximum Baseline score 0, worst post-baseline score missing | 0 | 0
  Maximum Baseline score 1, worst post-baseline score 0 | 3 | 0
  Maximum Baseline score 1, worst post-baseline score 1 | 59 | 5
  Maximum Baseline score 1, worst post-baseline score 2 | 21 | 1
  Maximum Baseline score 1, worst post-baseline score 3 | 6 | 2
  Maximum Baseline score 1, worst post-baseline score 4 | 1 | 0
  Maximum Baseline score 1, worst post-baseline score 5 | 1 | 0
  Maximum Baseline score 1, worst post-baseline score missing | 2 | 0
  Minimum Baseline score 0, worst post-baseline score 0 | 33 | 4
  Minimum Baseline score 0, worst post-baseline score 1 | 2 | 0
  Minimum Baseline score 0, worst post-baseline score 2 | 0 | 0
  Minimum Baseline score 0, worst post-baseline score 3 | 0 | 0
  Minimum Baseline score 0, worst post-baseline score 4 | 0 | 0
  Minimum Baseline score 0, worst post-baseline score 5 | 0 | 0
  Minimum Baseline score 0, worst post-baseline score missing | 0 | 0
  Minimum Baseline score 1, worst post-baseline score 0 | 19 | 2
  Minimum Baseline score 1, worst post-baseline score 1 | 71 | 5
  Minimum Baseline score 1, worst post-baseline score 2 | 1 | 1
  Minimum Baseline score 1, worst post-baseline score 3 | 0 | 0
  Minimum Baseline score 1, worst post-baseline score 4 | 0 | 0
  Minimum Baseline score 1, worst post-baseline score 5 | 0 | 0
  Minimum Baseline score 1, worst post-baseline score missing | 2 | 0

9. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG) Findings
Description: Electrocardiograms (ECG) was obtained after the participant has been in a semi-supine position for at least 5 min. ECG parameters included heart rate, PQ/PR duration, QRS and QT duration, QT Interval. Clinical significance was determined by the investigator. Number of participants with clinically significant abnormalities in 12-lead ECG were reported.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: Safety (SAF) analysis set included all participants who were administered any dose of any study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib | Tepotinib Monotherapy
Number analyzed (Participants) | 128 | 12
Participants | 21 | 1

10. Secondary Outcome: Combined Therapy: Objective Response According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1 Assessed by Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: Objective response was defined as percentage of participants with either a confirmed complete response (CR) or partial response (PR) from first administration of study treatment to first observation of progressive disease (PD). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
percentage of participants | 44.9 [34.8 to 55.3]

11. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Number of Participants With Confirmed Complete Response (CR) Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: Confirmed CR was defined as the disappearance of all evidence of target and non-target lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
Participants | 0

12. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Number of Participants With Confirmed Complete Response (CR) Assessed by Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: Confirmed CR was defined as the disappearance of all evidence of target and non-target lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
Participants | 1

13. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Duration of Response Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: DOR was defined for participants with objective response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: From first documented objective response to PD or death due to any cause, assessed approximately up to 42 months
Population: The primary analysis set for efficacy included all mFAS participants with advanced or metastatic EGFRm+ NSCLC and MET amplification, determined centrally by FISH (central TBx FISH testing [T+]). Here, Overall Number of Participants Analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 49
months | 8.5 [6.1 to NA] — Due to small number of events, upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not be derived.

14. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Duration of Response Assessed by Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 13
Time Frame: From first documented objective response to PD or death due to any cause, assessed approximately up to 42 months
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 44
months | 9.6 [7.1 to NA] — Due to small number of events, upper limit of 95% Confidence Interval from Kaplan-Meier survival curves could not be derived.

15. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Disease Control Rate Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: Disease control rate is defined as the percentage of participants with objective resposne (complete resposne [CR] or partial resposne [PR] or stable disease [SD]). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30 percent (%) reduction from baseline in the sum of the longest diameter (SLD) of all lesions. SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest SLD while on study. PD is defined as at least a 20 % increase in the SLD of target lesion, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
percentage of participants | 63.3 [52.9 to 72.8]

16. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Disease Control Rate Assessed by Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 15
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
percentage of participants | 64.3 [54.0 to 73.7]

17. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Progression-Free Survival (PFS) According to RECIST Version1.1 as Assessed by the Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: PFS was defined as the time is defined as the time from first administration of study treatment to the date of the first documentation of PD or death due to any cause within 126 days of the last tumor assessment, whichever occurs first. PD is defined as at least a 20 % increase in the SLD of target lesion, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first administration of study treatment to the date of the first documentation of PD or death due to any cause, assessed approximately up to 42 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
months | 5.6 [4.2 to 8.1]

18. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1as Assessed by the Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
months | 5.9 [4.2 to 8.5]

19. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Overall Survival in Participants With MET Amplification Determined Centrally by FISH
Description: Overall survival is defined as the time from first administration of study treatment to the date of death.
Time Frame: Time from first administration of study treatment to the date of death, assessed approximately up to 42 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 98
months | 17.8 [11.1 to NA] — Due to small number of events, upper limit of 95% confidence interval from Kaplan-Meier survival curves could not derive.

20. Secondary Outcome: Combined Therapy: Objective Response According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1as Assessed by Investigator in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: as for outcome 10
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: The secondary analysis set for efficacy included all mFAS participants with advanced or metastatic EGFRm+ NSCLC and MET amplification, determined centrally by liquid biopsy (LBx) test (L+).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
percentage of participants | 48.4 [30.2 to 66.9]

21. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Number of Participants With Confirmed Complete Response (CR) Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: Confirmed CR was defined as the disappearance of all evidence of target and non-target lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
Participants | 0

22. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Number of Participants With Confirmed Complete Response (CR) Assessed by Investigator in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: Confirmed CR was defined as the disappearance of all evidence of target and non-target lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
Participants | 0

23. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Duration of Response Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: as for outcome 13
Time Frame: From first documented objective response to PD or death due to any cause, assessed approximately up to 42 months
Population: The secondary analysis set for efficacy included all mFAS participants with advanced or metastatic EGFRm+ NSCLC and MET amplification, determined centrally by liquid biopsy (LBx) test (L+). Here, Overall Number of Participants Analyzed signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 17
months | 5.7 [2.9 to 15.4]

24. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Duration of Response Assessed by Investigator in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: as for outcome 13
Time Frame: From first documented objective response to PD or death due to any cause, assessed approximately up to 42 months
Population: as for outcome 23
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 15
months | 5.6 [2.9 to 9.6]

25. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Disease Control Rate Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: as for outcome 15
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
percentage of participants | 64.5 [45.4 to 80.8]

26. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Disease Control Rate Assessed by Investigator in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: as for outcome 15
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 20
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
percentage of participants | 67.7 [48.6 to 83.3]

27. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Progression-Free Survival (PFS) According to RECIST Version1.1 as Per Independent Review Committee in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
months | 5.5 [2.7 to 7.2]

28. Secondary Outcome: Combined Therapy ((Tepotinib + Osimertinib): Progression-Free Survival (PFS) According to RECIST Version1.1 as Assessed by the Investigator in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
months | 5.6 [4.2 to 7.0]

29. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Overall Survival in Participants With MET Amplification Determined Centrally by Blood-Based Next Generation Sequencing
Description: Overall survival is defined as the time from first administration of study treatment to the date of death.
Time Frame: Time from first administration of study treatment to the date of death, assessed approximately up to 42 months
Population: as for outcome 20
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 31
months | 13.7 [9.6 to NA] — Due to small number of events, upper limit of 95% confidence interval from Kaplan-Meier survival curves could not derive.

30. Secondary Outcome: Monotherapy (Tepotinib): Objective Response According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1as Per Investigator in Participants With MET Amplification Determined Centrally by Fluorescence in Situ Hybridization(FISH)
Description: as for outcome 2
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 12
percentage of participants | 8.3 [0.2 to 38.5]

31. Secondary Outcome: Monotherapy (Tepotinib): Number of Participants With Confirmed Complete Response (CR) Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: Confirmed CR was defined as the disappearance of all evidence of target and non-target lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 12
Participants | 0

32. Secondary Outcome: Monotherapy (Tepotinib): Number of Participants With Confirmed Complete Response (CR) Assessed by Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: Confirmed CR was defined as the disappearance of all evidence of target and non-target lesions.
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 12
Participants | 0

33. Secondary Outcome: Monotherapy (Tepotinib): Duration of Response Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 13
Time Frame: From first documented objective response to PD or death due to any cause, assessed approximately up to 42 months
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 1
months | 2.8 [NA to NA] — Insufficient number of participants with events, therefore 95% Confidence Interval could not be calculated.

34. Secondary Outcome: Monotherapy (Tepotinib): Duration of Response Assessed by Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 13
Time Frame: From first documented objective response to PD or death due to any cause, assessed approximately up to 42 months
Population: as for outcome 13
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 1
months | 2.8 [NA to NA] — Insufficient number of participants with events, therefore 95% Confidence Interval could not be calculated.

35. Secondary Outcome: Monotherapy (Tepotinib): Disease Control Rate Assessed by Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 15
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 12
percentage of participants | 25.0 [5.5 to 57.2]

36. Secondary Outcome: Monotherapy (Tepotinib): Disease Control Rate Assessed by Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 15
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 12
percentage of participants | 25.0 [5.5 to 57.2]

37. Secondary Outcome: Monotherapy (Tepotinib): Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1as Assessed by the Independent Review Committee in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 12
months | 2.7 [1.4 to 4.4]

38. Secondary Outcome: Monotherapy (Tepotinib): Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors(RECIST)Version1.1as Assessed by the Investigator in Participants With MET Amplification Determined Centrally by FISH
Description: as for outcome 17
Time Frame: as for outcome 17
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tepotinib Monotherapy
Number analyzed (Participants) | 12
months | 2.6 [1.4 to 4.4]

39. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Change From Baseline in European Quality Of Life 5-dimensions (EQ-5D-5L) Visual Analog Scale (VAS) at Safety Follow-up (42 Months)
Description: The EQ-5D-5L questionnaire is a generic measure of health status that provides a simple descriptive profile and a single index value. The EQ-5D-5L profile defines health in terms of mobility, self-care, usual activities, pain or discomfort, and anxiety or depression. Each dimension has five levels: 1: no problems, 2: slight problems, 3: moderate problems, 4: severe problems, and 5: extreme problems. The responses were used to derive overall score using a visual analog scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 was the worst health you can imagine and 100 was the best health you can imagine.
Time Frame: Baseline, safety follow-up (assessed up to 42 months)
Population: The primary analysis set for efficacy included all mFAS participants with advanced or metastatic EGFRm+ NSCLC and MET amplification, determined centrally by FISH (central TBx FISH testing [T+]). Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 41
score on a scale | -11 (21.7)

40. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life (EORTC QLQ-C30) Global Health Status) at Safety Follow-up (42 Months)
Description: EORTC QLQ-C30 was a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 15 domains: 1 global health status (GHS) scale, 5 functional scales (Physical, role, cognitive, emotional, social), and 9 symptom scales/items (Fatigue, nausea and vomiting, pain, dyspnea, sleep disturbance, appetite loss, constipation, diarrhea, financial impact). The EORTC QLQ-C30 GHS/QoL score ranged from 0 to 100; High score indicated better GHS/QoL. Score 0 represents: very poor physical condition and QoL. Score 100 represents: excellent overall physical condition and QoL.
Time Frame: Baseline, safety follow-up (up to 42 months)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 41
score on a scale | -6.5 (25.17)

41. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Change From Baseline in Health-Related Quality of Life as Assessed by Non-Small Cell Lung Cancer Symptom Assessment Questionnaire (NSCLC-SAQ) at Safety Follow-up (42 Months)
Description: NSCLC-SAQ was a question tool used to assess the overall quality of life (QoL) in cancer participants. It consisted of 5 domains: cough, pain, dyspnea, fatigue, and appetite. The NSCLC-SAQ score ranged from 0 to 20; High score indicated more severe NSCLC-related symptomatology. mains: cough, pain, dyspnea, fatigue, and appetite.
Time Frame: Baseline, safety follow-up (up to 42 months)
Population: as for outcome 39
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 42
score on a scale | 2.0 (4.26)

42. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t) of Tepotinib and Its Metabolites (MSC2571109A, MSC2571107A), Osimertinib and Its Metabolite AZD5104
Description: Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hours after tepotinib and Osimertinib administration at Day 1 of Cycle 1 and Day 15 of Cycle 1 (each Cycle is of 21 days) ]
Population: Pharmacokinetic analysis set included all FAS/SAF participants who have no important events affecting PK and provide at least one measurable post-dose concentration. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified timepoints for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*h/mL)
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 9
nanogram*hour per milliliter (ng*h/mL)
  Tepotinib: Cycle 1 Day 1 | 11600 (40.8)
  Tepotinib: Cycle 1 Day 15: number analyzed (Participants) | 6
  Tepotinib: Cycle 1 Day 15 | 26900 (47.1)
  MSC2571109A: Cycle 1 Day 1 | 2240 (40.0)
  MSC2571109A: Cycle 1 Day 15: number analyzed (Participants) | 6
  MSC2571109A: Cycle 1 Day 15 | 5160 (50.3)
  MSC2571107A: Cycle 1 Day 1 | 497 (292.6)
  MSC2571107A: Cycle 1 Day 15: number analyzed (Participants) | 5
  MSC2571107A: Cycle 1 Day 15 | 1180 (624.7)
  Osimertinib: Cycle 1 Day 1 | 9090 (168.9)
  Osimertinib: Cycle 1 Day 15: number analyzed (Participants) | 6
  Osimertinib: Cycle 1 Day 15 | 8710 (41.3)
  AZD5104: Cycle 1 Day 1 | 808 (424.6)
  AZD5104: Cycle 1 Day 15: number analyzed (Participants) | 6
  AZD5104: Cycle 1 Day 15 | 1010 (54.6)

43. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Maximum Observed Plasma Concentration (Cmax) of Tepotinib and Its Metabolites (MSC2571109A, MSC2571107A), Osimertinib and Its Metabolite AZD5104
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 42
Population: PK analysis set included all FAS/SAF participants who have no important events affecting PK and provide at least one measurable post-dose concentration. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "number analyzed" signifies those participants who were evaluable at specified timepoints for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 9
nanogram per milliliter (ng/mL)
  Tepotinib: Cycle 1 Day 1 | 660 (38.7)
  Tepotinib: Cycle 1 Day 15: number analyzed (Participants) | 6
  Tepotinib: Cycle 1 Day 15 | 1220 (45.1)
  MSC2571109A: Cycle 1 Day 1 | 167 (41.1)
  MSC2571109A: Cycle 1 Day 15: number analyzed (Participants) | 6
  MSC2571109A: Cycle 1 Day 15 | 274 (45.0)
  MSC2571107A: Cycle 1 Day 1 | 38.4 (26.57)
  MSC2571107A: Cycle 1 Day 15: number analyzed (Participants) | 5
  MSC2571107A: Cycle 1 Day 15 | 57.0 (27.19)
  Osimertinib: Cycle 1 Day 1 | 540 (144.6)
  Osimertinib: Cycle 1 Day 15: number analyzed (Participants) | 6
  Osimertinib: Cycle 1 Day 15 | 468 (51.2)
  AZD5104: Cycle 1 Day 1 | 43.6 (421.2)
  AZD5104: Cycle 1 Day 15: number analyzed (Participants) | 6
  AZD5104: Cycle 1 Day 15 | 50.9 (63.8)

44. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Time to Reach Maximum Observed Plasma Concentration (Tmax) of Tepotinib and Its Metabolites (MSC2571109A, MSC2571107A), Osimertinib and Its Metabolite AZD5104
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 42
Population: as for outcome 43
Measure: Median (Full Range); unit: hours
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 9
hours
  Tepotinib: Cycle 1 Day 1 | 23.97 [6.00 to 24.00]
  Tepotinib: Cycle 1 Day 15: number analyzed (Participants) | 6
  Tepotinib: Cycle 1 Day 15 | 5.13 [0.50 to 24.00]
  MSC2571109A: Cycle 1 Day 1 | 24.00 [12.00 to 24.00]
  MSC2571109A: Cycle 1 Day 15: number analyzed (Participants) | 6
  MSC2571109A: Cycle 1 Day 15 | 0.25 [0.00 to 24.77]
  MSC2571107A: Cycle 1 Day 1 | 24.00 [12.00 to 24.00]
  MSC2571107A: Cycle 1 Day 15: number analyzed (Participants) | 5
  MSC2571107A: Cycle 1 Day 15 | 24.00 [0.00 to 24.77]
  Osimertinib: Cycle 1 Day 1 | 6.00 [2.00 to 24.00]
  Osimertinib: Cycle 1 Day 15: number analyzed (Participants) | 6
  Osimertinib: Cycle 1 Day 15 | 5.00 [3.00 to 24.77]
  AZD5104: Cycle 1 Day 1 | 8.00 [1.50 to 24.00]
  AZD5104: Cycle 1 Day 15: number analyzed (Participants) | 6
  AZD5104: Cycle 1 Day 15 | 4.00 [0.00 to 24.77]

45. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Apparent Total Body Clearance (CL/f) of Tepotinib and Its Metabolites (MSC2571109A, MSC2571107A), Osimertinib and Its Metabolite AZD5104
Description: CL/f was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-t + Clast pred/Lambda Z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLQ) and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 42
Population: As per changes in planned analysis, the PK parameter (CL/f) was not assessed.
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 0

46. Secondary Outcome: Combined Therapy (Tepotinib + Osimertinib): Apparent Volume Of Distribution (Vz/F) of of Tepotinib and Its Metabolites (MSC2571109A, MSC2571107A), Osimertinib and Its Metabolite AZD5104
Description: Vz/f: the distribution of a study drug between plasma and the rest of the body after oral dosing. For single dose Vz/f = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-t + Clast pred/Lambda Z). Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z = the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 42
Population: As per changes in planned analysis, the PK parameter (Vz/f) was not assessed.
Arm/Group | Tepotinib + Osimertinib
Number analyzed (Participants) | 0

47. Secondary Outcome: Percentage of Participants With Resistant Mutations of the Epidermal Growth Factor Receptor (EGFR) Gene or Other Pathways as Assessed in Circulating Tumor Deoxyribonucleic Acid (ctDNA)
Description: Percentage of participants with resistant mutations of the EGFR gene or other pathways as assessed in ctDNA were reported.
Time Frame: From Day 1 of Cycle 3 up to end of treatment (14 days after last dose, approximately assessed up to 35.6 months) (each Cycle is for 21 days)
Population: As per changes in planned analysis, the data for mutation status in EGFR and other pathways in ctDNA at baseline and progression were not collected with the assay used to screen for MET amplification in ctDNA.
Arm/Group | Tepotinib + Osimertinib | Tepotinib Mono-therapy
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Time from first administration of study treatment up to data cutoff (approximately assessed up to 42 months)
Arm/Group | Tepotinib and Osimertinib | Tepotinib Mono-therapy
All-Cause Mortality (participants affected / at risk) | 59/128 | 7/12
Serious Adverse Events (participants affected / at risk) | 49/128 | 2/12
Other Adverse Events (participants affected / at risk) | 123/128 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tepotinib and Osimertinib (N=128) | Tepotinib Mono-therapy (N=12)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Disease progression (General disorders) | 5 (5) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cytolysis (Hepatobiliary disorders) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 5 (7) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Carbuncle (Infections and infestations) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 (2) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 3 (4) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral venous sinus thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tepotinib and Osimertinib (N=128) | Tepotinib Mono-therapy (N=12)
Anaemia (Blood and lymphatic system disorders) | 26 (31) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 3 (5) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (10) | 1 (1)
Extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (9) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 7 (7) | 0 (0)
Aerophagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 17 (18) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 69 (91) | 4 (6)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 7 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 36 (46) | 2 (4)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 25 (34) | 1 (1)
Asthenia (General disorders) | 13 (15) | 0 (0)
Chest pain (General disorders) | 2 (2) | 2 (2)
Fatigue (General disorders) | 11 (11) | 2 (2)
Non-cardiac chest pain (General disorders) | 4 (4) | 1 (1)
Oedema (General disorders) | 3 (3) | 1 (1)
Oedema peripheral (General disorders) | 60 (79) | 4 (6)
Pain (General disorders) | 3 (3) | 1 (1)
Pyrexia (General disorders) | 9 (10) | 1 (1)
COVID-19 (Infections and infestations) | 20 (27) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 29 (34) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (3) | 1 (1)
Urinary tract infection (Infections and infestations) | 7 (8) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 19 (22) | 2 (3)
Amylase increased (Investigations) | 15 (25) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 20 (23) | 1 (2)
Blood alkaline phosphatase increased (Investigations) | 10 (10) | 0 (0)
Blood bilirubin increased (Investigations) | 2 (2) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 7 (7) | 0 (0)
Blood creatinine increased (Investigations) | 16 (25) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 12 (15) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 3 (3)
Heart rate increased (Investigations) | 1 (2) | 1 (1)
Lipase increased (Investigations) | 18 (30) | 0 (0)
Lymphocyte count decreased (Investigations) | 7 (8) | 1 (1)
Neutrophil count decreased (Investigations) | 8 (15) | 1 (1)
Platelet count decreased (Investigations) | 14 (20) | 0 (0)
Red blood cells urine positive (Investigations) | 0 (0) | 1 (1)
Urine bilirubin increased (Investigations) | 0 (0) | 1 (1)
Urine ketone body present (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 18 (19) | 1 (1)
Weight increased (Investigations) | 3 (4) | 1 (1)
White blood cell count decreased (Investigations) | 7 (15) | 1 (1)
White blood cells urine positive (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 30 (35) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (9) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 35 (42) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 19 (25) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 8 (16) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 12 (19) | 1 (1)
Hypoproteinaemia (Metabolism and nutrition disorders) | 6 (6) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (9) | 2 (2)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (5) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 8 (8) | 1 (1)
Proteinuria (Renal and urinary disorders) | 4 (5) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 (18) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 1 (1)
Vasomotor rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vocal cord fixation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 14 (15) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT03940703/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-04): https://cdn.clinicaltrials.gov/large-docs/03/NCT03940703/SAP_001.pdf